CLINICAL TRIAL: NCT01655329
Title: Reader Study to Demonstrate That Use of ClearRead Confirm is Superior to the Use Standard AP/PA X-ray Image. AP Stands for Antero-Posterior. PA Stands for Postero-anterior.
Brief Title: Reader Study to Demonstrate That Use of ClearRead Confirm is Superior to the Use Standard AP/PA X-ray Image
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: Riverain Technologies (Industry)
Responsible Party: Principal Investigator, Matthew T. Freedman, MD, Associate Professor Oncology, Georgetown University
Other Study IDs: MF 2012-1
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: Catheters, With or Without Malposition; Image Interpretation, Computer Assisted
Keywords: Image Processing; tubes; lines; catheters; wires; Bedside; chest; radiographs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard chest radiographs: The radiologists will be viewing two groups of chest images. The first group are standard chest radiographs.
- Modified chest radiographs: This group of chest radiographs will be presented with the modified image. The modified image is intended to increase the visibility of tubes, lines and wires on chest radiographs

SUMMARY:
This is a study to determine whether or not a new type of software is, or is not, of benefit. The software, ClearRead Confirm, is designed to enhance the ability of radiologists to detect tubes, lines and wires that may be placed within a patients chest. These types of devices are commonly used for very sick patients in intensive care units and are also used following surgery and in the treatment of cancer. This study will test radiologist's detection of the tips of these devices comparing the results with standard chest radiographs and the the modified chest radiographs. The primary interest is in the time used to interpret the radiograph. We will determine if there is any change in accuracy of detection.

DETAILED DESCRIPTION:
Primary hypothesis: the amount of time used for the interpretation of these radiographs will not change. (null hypothesis)

Secondary hypothesis: there will be no change in the accuracy of the detection of the tips of venous catheters and tubes transiting the esophagus. (null hypothesis)

ELIGIBILITY:
Inclusion Criteria:

* For the radiologists, they must in in active practice of community radiology (non-university sites).
* For the cases, they must be patients who have a tube, line, or wire in their chest. A small number of completely normal bedside chest radiographs will be included.

Exclusion Criteria:

* For radiologists: Not in active practice. Working in a university hospital.
* For cases: children. Do not meet image quality criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are two populations: the radiologists and the cases they will review. For cases, these are sequential cases selected by database search using defined search criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Freedman, MD, MBA, Principal Investigator — Georgetown University; Shih-Chung Ben Lo, Ph.D., Study Director — Georgetown University
Locations (1):
- Georgetown University Medical Center, Suite 603, 2115 Wisconsin Ave, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten Board Certified radiologists practicing in community (non-university) practice were recruited from the Washington, DC, - Baltimore, MD, Metropolitan region. Recruitment was by email and phone calls to prior participants in our studies and to other radiologists that they referred us to. Recruitment April, 2012 through September, 2012
Pre-assignment Details: 54 cases were used to train the radiologists on the use of the data recording computer and to make them familiar with the appearance of the processed chest radiographs. These cases were not used in the test of reader performance.
Groups:
- Chest Radiographs: The radiologists will be viewing two groups of chest images. The first group are standard chest radiographs. The second group are the processed images. These radiographs were randomly placed into two groups. The radiologists were randomly placed in two groups. Each of these two groups interpreted half of the standard chest radiograph without processing and half with the special processing. The other group of radiologists interpreted the other half of the normal and the other half of the processed images. The radiologists reviewed each radiograph using one or the alternate presentation
Period: Overall Study
Arm/Group | Chest Radiographs
Started | 10 (The same 10 radiologists are interpreting images in both arms.)
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Board Certified Radiologists
Groups:
- Radiologists: Board Certified Radiologists
Arm/Group | Radiologists
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  female | 3
  male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Time for Completion of Tasks
Description: Time for completion of tasks of identifying the tips of tubes, lines, and wires. Outlying values are excluded from the calculation of the mean values and standard errors. Outlying values were defined as those more than three standard deviations from the mean time.
Time Frame: 8 hours
Population: Each radiologist interpreted only half (158) chest radiographs. All of the radiographs were interpreted by a combination of the 10 radiologist participants.
Measure: Mean (Standard Error); unit: seconds
Units Other Than Participants: chest radiographs
Groups:
- Standard Chest Radiographs: The radiologists will be viewing two groups of chest images. The first group are standard chest radiographs. The second group are the processed images. These radiographs were randomly placed into two groups. The radiologists were randomly placed in two groups. Each of these two groups interpreted half of the standard chest radiograph without processing and half with the special processing. The other group of radiologists interpreted the other half of the normal and the other half of the processed images.
- Modified Chest Radiographs: This group of chest radiographs will be presented with the modified image. The modified image is intended to increase the visibility of tubes, lines and wires on chest radiographs. Each radiologist interpreted half the images as conventional images and half as processed images.
Arm/Group | Standard Chest Radiographs | Modified Chest Radiographs
Number analyzed (Participants) | 10 | 10
Number analyzed (chest radiographs) | 334 | 334
seconds | 27.68 (3.32) [21.04 to 34.24] | 22.90 (3.32) [16.34 to 29.46]

2. Primary Outcome: Accuracy in Detecting the Tips of Tubes, Lines, and Wires.
Description: Measurement of accuracy in determining the location of the tips of nasogastric tubes (NG) (various types of nasogastric tubes combined) and of the tips of venous catheters (various types of venous catheters combined), compared to the determination of the expert panel. Measure is the distance from the median location determined by five experts in chest radiology.
Time Frame: 8 hours
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Standard Chest Radiographs | Modified Chest Radiographs
Number analyzed (Participants) | 10 | 10
centimeters
  NG tubes distance in centimeters vs experts | 3.62 (0.79) [NA to NA] | 3.96 (0.78) [NA to NA]
  Venous catheters distance in centimeters | 3.49 (0.52) [NA to NA] | 3.14 (0.52) [NA to NA]

3. Other Pre Specified Outcome: Likert-Like
Description: Following the viewing of the test radiographs, the radiologists were asked a series of questions of overall preference. On this scale, 1 indicates strong disagreement, 5 indicates strongly agree. Ten statements were used. Note that a low value for the standard image is equivalent to a high value for the modified image.
Time Frame: 10 minutes
Population: All 10 radiologist participants participated
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Reading Time Estimate by Radiologists: The modified image will reduce reading time.
- Pleural Drain Visibility: Pleural drains are easier to see on the standard image.
- Venous Catheters: Venous catheters easier to see on modified image
- Cardiac Related Wires: Cardiac related wires are easier to see on the standard image
- Overall Image Quality: Overall image quality is superior on the standard image
- Image Quality Radioopaque Regions: Image quality in the opaque image areas is superior on the confirm image
- Confidence on Line Placement: The modified image increased my confidence with respect to line placement
- Need for Window/Level Manipulation: The standard image required less window/level manipulation
- Confidence on Tube Placement: The confirm image increases my confidence with respect to tube placement.
Arm/Group | Reading Time Estimate by Radiologists | Pleural Drain Visibility | Venous Catheters | Cardiac Related Wires | Overall Image Quality | Image Quality Radioopaque Regions | Confidence on Line Placement | Need for Window/Level Manipulation | Confidence on Tube Placement
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
units on a scale | 3.9 (0.99) | 2.4 (0.97) | 4.5 (0.71) | 2.7 (1.34) | 2.5 (1.08) | 2.9 (1.29) | 4.1 (1.29) | 1.6 (1.26) | 4.4 (0.70)

ADVERSE EVENTS:
Description: Injuries to radiologists during study. No systematic assessment was made of injuries to the radiologists.
Arm/Group | Radiologists
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days